CLINICAL TRIAL: NCT03518034
Title: Testosterone Replacement Therapy for Assessment of Long-term Vascular Events and Efficacy ResponSE in Hypogonadal Men (TRAVERSE) Study
Brief Title: A Study to Evaluate the Effect of Testosterone Replacement Therapy (TRT) on the Incidence of Major Adverse Cardiovascular Events (MACE) and Efficacy Measures in Hypogonadal Men
Acronym: TRAVERSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Endo Pharmaceuticals (Industry); Acerus Pharmaceuticals Corporation (Industry); Allergan Sales, LLC (Industry); Upsher-Smith Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-100
Record Dates: First submitted 2018-05-03; First posted 2018-05-08 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Hypogonadism; Cardiovascular Diseases
Keywords: hypogonadism; cardiovascular (CV) disease; AndroGel; testosterone replacement therapy (TRT)
MeSH Terms: conditions — Hypogonadism; Cardiovascular Diseases; Disease | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AndroGel 1.62% (Active Comparator): Participants receive topical testosterone starting with a 40.5 mg dose (2 pump actuations) of the study drug once daily (OD). Participants may receive a dose in the range of 20.25 mg (1 actuation) to 101.25 mg (5 actuations) in 20.25 mg increments during the course of the study if titrations are necessary.
  Interventions: Drug: AndroGel®
- Placebo (Placebo Comparator): Participants receive matching placebo OD.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AndroGel® — testosterone administered topically
  Arms: AndroGel 1.62%
Drug: Placebo — placebo administered topically
  Arms: Placebo

SUMMARY:
This is a double-blinded and placebo-controlled study of topical testosterone replacement therapy (TRT) in symptomatic hypogonadal men with pre-existing cardiovascular disease (CVD) or increased risk for CVD.

ELIGIBILITY:
Inclusion Criteria:

* Men between 45 and 80 years age
* Participants with low serum testosterone concentrations (< 300 ng/dL) who exhibit at least one sign or symptom of hypogonadism and have evidence of cardiovascular (CV) disease or are at an increased risk for CV disease.

Exclusion Criteria:

* Participants with congenital or acquired hypogonadism for whom long-term therapy with placebo would not be medically appropriate
* Participants with prostate specific antigen (PSA) > 3.0 ng/mL (or 1.5 if on 5-alpha reductase inhibitors)
* Participants who have been treated with testosterone in the past 6 months and for whom testosterone therapy is contraindicated
* Confirmed testosterone < 100 ng/dL
* Body Mass Index (BMI) > 50
* Hemoglobin A1c (HbA1C) > 11%
* Hematocrit (Hct) > 50%
* Estimated Glomerular Filtration Rate (eGFR) < 30 ml/min
* History of deep vein thrombosis or pulmonary embolism or prostate cancer or heart failure (Class III and IV).

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5246 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (384):
- United States (379):
  - Wright Clinical Research, LLC /ID# 210864, Alabaster, Alabama
  - Simon-Williamson Clinic /ID# 210249, Birmingham, Alabama
  - Alabama Clinical Therapeutics /ID# 202982, Birmingham, Alabama
  - Cahaba Research, Inc. /ID# 167928, Birmingham, Alabama
  - Atlanta VAHCS /ID# 170318, Decatur, Alabama
  - G & L Research, LLC /ID# 170365, Foley, Alabama
  - Fundamental Research /ID# 170504, Gulf Shores, Alabama
  - Urology Centers of Alabama /ID# 206197, Homewood, Alabama
  - Longwood Research /ID# 201754, Huntsville, Alabama
  - Medical Affiliated Research Center, Inc. /ID# 170569, Huntsville, Alabama
  - Mostellar Medical Center /ID# 170329, Mobile, Alabama
  - Terence T. Hart, MD /ID# 201561, Tuscumbia, Alabama
  - Alaska Urological Institute /ID# 167894, Anchorage, Alaska
  - Synexus Clinical Research US, INC /ID# 170530, Chandler, Arizona
  - Fountain Hills Family Practice P.C /ID# 170419, Fountain Hills, Arizona
  - Horizon Clinical Research Asoc /ID# 202937, Gilbert, Arizona
  - Lenzmeier Family Medicine /ID# 202945, Glendale, Arizona
  - Synexus - Desert Clinical Research /ID# 170428, Mesa, Arizona
  - Phoenix Medical Group, PC /ID# 170516, Peoria, Arizona
  - Phoenix VA Health Care System /ID# 167968, Phoenix, Arizona
  - Elite Clinical Studies, LLC /ID# 168058, Phoenix, Arizona
  - Family Practice Specialists /ID# 167859, Phoenix, Arizona
  - Central Phoenix Medical Clinic /ID# 170333, Phoenix, Arizona
  - Tatum Highlands Medical Assoc /ID# 208277, Phoenix, Arizona
  - Fiel Family & Sports Medicine /ID# 203034, Tempe, Arizona
  - Arizona Research Assoc /ID# 170421, Tucson, Arizona
  - Quality of Life Medical & Research Center /ID# 167915, Tucson, Arizona
  - Southern Arizona VA Health Care System /ID# 167600, Tucson, Arizona
  - Verde Valley Medical Center /ID# 202955, Tucson, Arizona
  - Eclipse Clinical Research /ID# 170381, Tucson, Arizona
  - B.G. Clinical Research Center, LLC /ID# 170461, Little Rock, Arkansas
  - Preferred Research Partners /ID# 170539, Little Rock, Arkansas
  - Applied Research Center of Arkansas /ID# 170487, Little Rock, Arkansas
  - Pacific Oaks Medical Group /ID# 170540, Beverly Hills, California
  - West Coast Research LLC /ID# 167903, Dublin, California
  - Diagnamics Inc. /ID# 205836, Encinitas, California
  - Cedars Sinai Medical Group /ID# 170383, Encino, California
  - St. Jude Hospital Yorba Linda /ID# 170437, Fullerton, California
  - Arizona Internal Medicine Specialists, LLC- Glendale /ID# 203011, Glendale, California
  - Allied Clinical Research /ID# 170519, Gold River, California
  - Marvel Clinical Research, LLC /ID# 170324, Huntington Beach, California
  - Irvine Center for Clinical Research /ID# 170368, Irvine, California
  - San Diego Clinical Trials /ID# 170468, La Mesa, California
  - TriWest Research Associates- La Mesa /ID# 170498, La Mesa, California
  - Clinical Trials Research /ID# 210862, Lincoln, California
  - Torrance Clinical Research Institute, Inc. /ID# 170307, Lomita, California
  - VA Long Beach Healthcare System /ID# 170374, Long Beach, California
  - Tower Urology /ID# 170330, Los Angeles, California
  - Facey Medical Foundation /ID# 203004, Mission Hills, California
  - Catalina Research Institute, LLC /ID# 170501, Montclair, California
  - NewportNativeMD, Inc. /ID# 168110, Newport Beach, California
  - Velocity Clinical Research, Inc. /ID# 168115, North Hollywood, California
  - Valley Clinical Trials - Northridge Location /ID# 201587, Northridge, California
  - Valley Renal Medical Group /ID# 170587, Northridge, California
  - Diabetes Associates Medical Group /ID# 170499, Orange, California
  - Desert Oasis Healthcare /ID# 170841, Palm Springs, California
  - Saviers Medical Group /ID# 170327, Port Hueneme, California
  - Stanford University /ID# 167595, Redwood City, California
  - Center for Clinical Trials of Sacramento, Inc. /ID# 168108, Sacramento, California
  - Integrated Research Center, Inc. /ID# 170391, San Diego, California
  - Ritchken & First MD's /ID# 201341, San Diego, California
  - San Diego Sexual Medicine /ID# 170457, San Diego, California
  - VA San Diego Healthcare System /ID# 168252, San Diego, California
  - Syrentis Clinical Research /ID# 168056, Santa Ana, California
  - Care Access Research /ID# 167916, Santa Clarita, California
  - Encompass Clinical Research /ID# 202203, Spring Valley, California
  - St. Joseph's Medical Associate /ID# 170424, Stockton, California
  - Olive View UCLA Medical Center /ID# 206131, Sylmar, California
  - Millennium Clinical Trials /ID# 210695, Thousand Oaks, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center /ID# 170400, Torrance, California
  - Bayview Research Group LLC /ID# 203036, Valley Village, California
  - Anthony Mills, MD, Inc. /ID# 170571, West Hollywood, California
  - Lynn Institute of Denver /ID# 170312, Aurora, Colorado
  - Lynn Institute of Colorado Springs South /ID# 168231, Colorado Springs, Colorado
  - Lynn Institute of the Rockies /ID# 170477, Colorado Springs, Colorado
  - Urology Associates of Colorado /ID# 170484, Englewood, Colorado
  - New West Physicians /ID# 203032, Golden, Colorado
  - Advanced Urology, PLLC dba Colorado Clinical Research /ID# 170406, Lakewood, Colorado
  - Aventura Heart Center /ID# 170354, Aventura, Florida
  - MB Clinical Research /ID# 202970, Boca Raton, Florida
  - Imagine Research of Palm Beach County /ID# 212140, Boynton Beach, Florida
  - Helix Biomedics, LLC /ID# 202310, Boynton Beach, Florida
  - Meridien Research Inc. - Brooksville /ID# 170556, Brooksville, Florida
  - Innovative Research of West Florida /ID# 170360, Clearwater, Florida
  - Tampa Bay Medical Res, Inc /ID# 170512, Clearwater, Florida
  - ALL Medical Research /ID# 170493, Cooper City, Florida
  - Century Clinical Research, Inc /ID# 167597, Daytona Beach, Florida
  - Seidman Clinical Trials,Delray /ID# 170418, Delray Beach, Florida
  - S&W Clinical Research /ID# 170311, Fort Lauderdale, Florida
  - Invesclinic, U.S., LLC /ID# 202553, Fort Lauderdale, Florida
  - The Center for Diabetes and Endocrine Care /ID# 170373, Fort Lauderdale, Florida
  - University of Florida - Hull Rd /ID# 170518, Gainesville, Florida
  - Malcom Randall VAMC /ID# 170645, Gainesville, Florida
  - Indago Research and Health Cen /ID# 170420, Hialeah, Florida
  - South Florida Research Solutions, LLC /ID# 167972, Hollywood, Florida
  - The University of Florida Heal /ID# 170450, Jacksonville, Florida
  - Jacksonville Center for Clinical Research /ID# 170446, Jacksonville, Florida
  - Solutions Through Adv Rch /ID# 201590, Jacksonville, Florida
  - Care Partners Clinical Research /ID# 202520, Jacksonville, Florida
  - Health Awareness, Inc - Port St Lucie /ID# 170507, Jupiter, Florida
  - Meridien Research /ID# 167846, Lakeland, Florida
  - South Florida Wellness & Clinic /ID# 170510, Margate, Florida
  - Panax Clinical Research /ID# 170525, Miami, Florida
  - Pharmax Research Clinic /ID# 170403, Miami, Florida
  - APF Research, LLC. /ID# 170412, Miami, Florida
  - Well Pharma Medical Research /ID# 170337, Miami, Florida
  - Advanced Pharma CR, LLC /ID# 167840, Miami, Florida
  - Applemed Research Inc. /ID# 170364, Miami, Florida
  - New Horizon Research Center /ID# 170574, Miami, Florida
  - Future Care Solution LLc /ID# 170361, Miami, Florida
  - Care Research center Inc. /ID# 167924, Miami, Florida
  - Office of Francisco G Miranda, /ID# 203184, Miami, Florida
  - Floridian Research Institute LLC /ID# 167882, Miami, Florida
  - International Research Associates, LLC /ID# 170543, Miami, Florida
  - International Research Associates, LLC /ID# 170563, Miami, Florida
  - Quantum Clinical Trials /ID# 224233, Miami Beach, Florida
  - Meridian International Research, Inc. /ID# 202975, Miami Lakes, Florida
  - Bravo Health Care Center /ID# 202201, North Bay Village, Florida
  - Harmony Clinical Research, Inc. /ID# 201816, North Miami Beach, Florida
  - Endocrine Associates of Florida, P.A. /ID# 167839, Ocoee, Florida
  - Sensible Healthcare /ID# 170402, Ocoee, Florida
  - Omega Research Group /ID# 170340, Orlando, Florida
  - IMIC Inc. Medical Research /ID# 167899, Palmetto Bay, Florida
  - South Broward Research /ID# 170480, Pembroke Pines, Florida
  - DBC Research USA /ID# 170332, Pembroke Pines, Florida
  - Synexus Clinical Research US, Inc /ID# 209955, Pinellas Park, Florida
  - DMI Research, Inc. /ID# 170893, Pinellas Park, Florida
  - Clinical Research Center FL /ID# 202979, Pompano Beach, Florida
  - St. Johns Center /ID# 212654, Ponte Vedra, Florida
  - Charlotte Heart & Vascular Institute /ID# 202965, Port Charlotte, Florida
  - Accel Research Sites - St Petersburg Clinical Research Unit /ID# 170370, St. Petersburg, Florida
  - Professional Health Care of Pinellas /ID# 167895, St. Petersburg, Florida
  - Advance Medical Research /ID# 170532, St. Petersburg, Florida
  - Precision Clinical Research /ID# 170469, Sunrise, Florida
  - DBC Research Corp /ID# 170435, Tamarac, Florida
  - Accel Research Sites - Tampa Clinical Research Unit /ID# 170377, Tampa, Florida
  - Winter Park Urology Center/Charter Research /ID# 210542, Winter Park, Florida
  - Atlanta Vascular Research Foundation - Atlanta Clinical Research Centers /ID# 170894, Atlanta, Georgia
  - Masters of Clinical Research, Inc. /ID# 167950, Augusta, Georgia
  - Endocrine Consustants Research /ID# 168147, Columbus, Georgia
  - Physicians Research Associates, LLC /ID# 170313, Lawrenceville, Georgia
  - Atlanta Center for Clinical Research /ID# 202984, Roswell, Georgia
  - Meridian Clinical Research LLC /ID# 167854, Savannah, Georgia
  - Meridian Clinical Research LLC /ID# 170548, Savannah, Georgia
  - Herman Clinical Research, LLC /ID# 170474, Suwanee, Georgia
  - North Georgia Clinical Research /ID# 170467, Woodstock, Georgia
  - East-West Medical Research Institute /ID# 202959, Honolulu, Hawaii
  - Institute of Arthritis Research /ID# 170495, Idaho Falls, Idaho
  - Solaris Clinical Research /ID# 202936, Meridian, Idaho
  - Biofortis, Inc. /ID# 167856, Addison, Illinois
  - Synexus Clinical Research US, Inc /ID# 209956, Chicago, Illinois
  - Chicago Clinical Research Institute, Inc /ID# 203190, Chicago, Illinois
  - Loretto Hospital.Affnity Clinical Research Institute /ID# 207262, Chicago, Illinois
  - Midwest Endocrinology /ID# 202992, Crystal Lake, Illinois
  - Dupage Medical Group /ID# 219039, Evergreen Park, Illinois
  - Pharmakon Inc /ID# 206149, Evergreen Park, Illinois
  - Clinical Investigation Specialists, Inc. /ID# 170631, Gurnee, Illinois
  - Edward Hines Jr. VA Hospital /ID# 167944, Hines, Illinois
  - Koch Family Medicine SC /ID# 202205, Morton, Illinois
  - Affinity Health /ID# 202552, Oak Brook, Illinois
  - American Health Network of IN, LLC (Avon) /ID# 170359, Avon, Indiana
  - Investigators Research Group, LLC /ID# 170557, Brownsburg, Indiana
  - Investigative Clinical Research of Indiana, LLC /ID# 170473, Elwood, Indiana
  - Deaconess Clinic Downtown /ID# 167855, Evansville, Indiana
  - Clinical Research Advantage, Inc. /ID# 170656, Evansville, Indiana
  - MediSphere Medical Research Center /ID# 170317, Evansville, Indiana
  - American Health Network of IN, LLC (Avon) /ID# 170483, Franklin, Indiana
  - Richard L. Roudebush VA Medical Center /ID# 203020, Indianapolis, Indiana
  - Urology of Indiana - Naab Road /ID# 203469, Indianapolis, Indiana
  - First Urology,PSC /ID# 167719, Jeffersonville, Indiana
  - LaPorte County Institute for Clinical Research, Inc. /ID# 170331, Michigan City, Indiana
  - American Health Network of Indiana, LLC /ID# 170578, Muncie, Indiana
  - West Broadway Clinic /ID# 202204, Council Bluffs, Iowa
  - Iowa Diabetes and Endocrinology Research Center /ID# 170462, West Des Moines, Iowa
  - The Iowa Clinic, PC /ID# 202986, West Des Moines, Iowa
  - Heartland Research Associates, LLC /ID# 203031, El Dorado, Kansas
  - Alliance for Multispecialty Research (AMR) - Wichita West /ID# 170415, Wichita, Kansas
  - Drs. Borders, Hood, and Assoc /ID# 170536, Lexington, Kentucky
  - The Research Grp of Lexington /ID# 202900, Lexington, Kentucky
  - University of Louisville /ID# 170607, Louisville, Kentucky
  - Research Integrity, LLC /ID# 168264, Owensboro, Kentucky
  - Alexandria Cardiology Clinic /ID# 170463, Alexandria, Louisiana
  - Centex Studies, Inc /ID# 170416, Lake Charles, Louisiana
  - Tandem Clinical Research, LLC /ID# 206203, Marrero, Louisiana
  - Barnum Internal Medicine /ID# 170343, Natchitoches, Louisiana
  - Tulane School of Medicine /ID# 170472, New Orleans, Louisiana
  - Maryland Cardiovascular Specialists /ID# 168057, Baltimore, Maryland
  - Johns Hopkins University /ID# 203006, Baltimore, Maryland
  - Centennial Medical Group /ID# 170568, Elkridge, Maryland
  - NECCR PrimaCare Research, LLC /ID# 170326, Fall River, Massachusetts
  - Oakland Medical Research /ID# 170389, Troy, Michigan
  - Arcturus Healthcare, PLC, Troy Internal Medicine Research Division /ID# 170431, Troy, Michigan
  - Olive Branch Family Med Ctr /ID# 170409, Olive Branch, Mississippi
  - David M. Headley, MD, P.A. /ID# 205428, Port Gibson, Mississippi
  - West Florissant Internists /ID# 170314, Bridgeton, Missouri
  - Med Research One /ID# 167923, Florissant, Missouri
  - Mercy Clinic Endocrinology, LLC /ID# 170367, Springfield, Missouri
  - St. Louis University /ID# 170531, St Louis, Missouri
  - Synexus Clinical Research US, Inc. /ID# 209957, St Louis, Missouri
  - Montana Medical Research /ID# 170579, Missoula, Montana
  - Skyline Medical Center /ID# 168234, Elkhorn, Nebraska
  - VA Nebraska-Western Iowa Health Care System /ID# 167892, Omaha, Nebraska
  - Heartland Clinical Research /ID# 170541, Omaha, Nebraska
  - Meridian Clinical Research, LLC - Omaha /ID# 167836, Omaha, Nebraska
  - Clinical Research Advantage, Inc. /ID# 202966, Omaha, Nebraska
  - Synexus Clinical Research US Inc /ID# 170560, Omaha, Nebraska
  - Alas Science Clinical Research /ID# 170352, Henderson, Nevada
  - Synexus Clinical Research US, Inc. /ID# 210232, Henderson, Nevada
  - AB Clinical Trials /ID# 170612, Las Vegas, Nevada
  - Clinical Research of So Nevada /ID# 167594, Las Vegas, Nevada
  - Advanced Biomedical Research of America /ID# 202202, Las Vegas, Nevada
  - Palm Research Center, Inc. /ID# 168224, Las Vegas, Nevada
  - Sheldon Freedman MD, ltd /ID# 170434, Las Vegas, Nevada
  - Allied Clinical Research /ID# 210859, Reno, Nevada
  - Internal Medicine Associates /ID# 170538, Bridgeton, New Jersey
  - Medicor Cardiology /ID# 170436, Bridgewater, New Jersey
  - Cooper Health System /ID# 170417, Camden, New Jersey
  - Union Square Medical Associates,PC /ID# 170346, Elizabeth, New Jersey
  - IMA Clinical research- Warren /ID# 170452, Warren Township, New Jersey
  - NM Clinical Research & Osteoporosis Center, Inc /ID# 170386, Albuquerque, New Mexico
  - Albany Stratton VA Medical Center /ID# 167862, Albany, New York
  - NY Total Medical Care, PC /ID# 170423, Brooklyn, New York
  - AccuMed Research Associates /ID# 202200, Garden City, New York
  - Office of Bruce R. Gilbert, MD /ID# 202963, Great Neck, New York
  - Synexus Clinical Research US, Inc. /ID# 210293, Jamaica, New York
  - Mid Hudson Medical Research, PLLC /ID# 170511, New Windsor, New York
  - Manhattan Medical Research /ID# 167956, New York, New York
  - DiGiovanna Institute for Medical Education & Research /ID# 170613, North Massapequa, New York
  - Premier Medical Group of the Hudson Valley PC /ID# 170456, Poughkeepsie, New York
  - Endocrine Assc Long Island PC /ID# 170425, Smithtown, New York
  - James J. Peters VA Medical Center /ID# 202980, The Bronx, New York
  - Randolph Health Internal Medicine /ID# 168227, Asheboro, North Carolina
  - OnSite Clinical Solutions, LLC - Hickory /ID# 170449, Charlotte, North Carolina
  - PMG Research of Charlotte /ID# 202985, Charlotte, North Carolina
  - OnSite Clinical Solutions, LLC /ID# 170349, Charlotte, North Carolina
  - OnSite Clinical Solutions, LLC /ID# 170634, Charlotte, North Carolina
  - Rapha Institute for Clinical Research /ID# 170362, Fayetteville, North Carolina
  - Bland Clinic, PA /ID# 204943, Greensboro, North Carolina
  - Medication Management, LLC /ID# 205260, Greensboro, North Carolina
  - Triad Clinical Trials /ID# 170376, Greensboro, North Carolina
  - OnSite Clinical Solutions, LLC - Hickory /ID# 202968, Hickory, North Carolina
  - Northstate Clinical Research /ID# 170414, Lenoir, North Carolina
  - PMG Research of Piedmont Healthcare /ID# 170341, Mooresville, North Carolina
  - Carteret Medical Group LLC /ID# 170771, Morehead City, North Carolina
  - Diabetes & Endocrinology Consultants /ID# 201589, Morehead City, North Carolina
  - Family Medical Associates of Raleigh /ID# 203979, Raleigh, North Carolina
  - Goshen Medical Center - Vineland /ID# 170342, Whiteville, North Carolina
  - PMG Research of Wilmington LLC /ID# 170492, Wilmington, North Carolina
  - Synexus Clinical Research, Inc /ID# 202976, Akron, Ohio
  - Velocity Clinical Research /ID# 170460, Blue Ash, Ohio
  - Diabetes and Endocrinology Associates of Stark County Inc /ID# 170356, Canton, Ohio
  - Gabrail Cancer Center Research /ID# 170533, Canton, Ohio
  - Cincinnati Veterans Affairs Medical Center /ID# 170385, Cincinnati, Ohio
  - Synexus Research Cincinnati /ID# 209958, Cincinnati, Ohio
  - Velocity clinical research /ID# 170513, Cleveland, Ohio
  - Endocrinology Associates, Inc. /ID# 168113, Columbus, Ohio
  - Synexus Clinical Research US, Inc. /ID# 210234, Columbus, Ohio
  - The Ohio State University Wexner Medical Center - Department of Urology /ID# 170551, Columbus, Ohio
  - Aventiv Research Columbus /ID# 170338, Columbus, Ohio
  - Optimed Research, Ltd. /ID# 168111, Columbus, Ohio
  - PriMed Clinical Research /ID# 170310, Dayton, Ohio
  - Dayton VA Medical Center /ID# 168251, Dayton, Ohio
  - WVVA Healthcare Alliance dba. /ID# 168246, Lewisburg, Ohio
  - Awasty Research Network, LLC /ID# 210860, Marion, Ohio
  - Advanced Medical Research /ID# 170488, Maumee, Ohio
  - Mercy Health St. Vincent Medical Center, LLC, Clinical Research Office /ID# 203035, Toledo, Ohio
  - Alliance for Multispecialty Research- Norman /ID# 170581, Norman, Oklahoma
  - IPS Research Company /ID# 168117, Oklahoma City, Oklahoma
  - Lynn Health Science Institute East /ID# 170497, Oklahoma City, Oklahoma
  - Lynn Health Science Institute (LHSI) /ID# 202973, Oklahoma City, Oklahoma
  - MidLantic Urology /ID# 170351, Bala-Cynwyd, Pennsylvania
  - Heritage Valley Medical Group /ID# 170387, Beaver, Pennsylvania
  - Feasterville Family Health Care Center /ID# 168235, Feasterville, Pennsylvania
  - Indiana-Armstrong Endocrinolgy /ID# 168249, Indiana, Pennsylvania
  - Richard M Kastelic, MD and Ass /ID# 170382, Johnstown, Pennsylvania
  - Family Medical Associates /ID# 170396, Levittown, Pennsylvania
  - Founders Research Corp /ID# 170610, Philadelphia, Pennsylvania
  - Allegheny Health Network /ID# 210544, Pittsburgh, Pennsylvania
  - Pittsburgh VA Medical Center-University Drive /ID# 205837, Pittsburgh, Pennsylvania
  - SFM Clinical Trials /ID# 168250, Scotland, Pennsylvania
  - Frontier Clinical Research, LLC - Scottdale /ID# 167864, Scottdale, Pennsylvania
  - Frontier Clinical Research /ID# 167842, Smithfield, Pennsylvania
  - Ocean State Clin Rese Part,LLC /ID# 170547, Lincoln, Rhode Island
  - Synexus Clinical Research US, Inc. /ID# 210230, Anderson, South Carolina
  - Synexus Clinical Research US, Inc. /ID# 210228, Anderson, South Carolina
  - Medical Research South, LLC /ID# 203068, Charleston, South Carolina
  - Synexus Clinical Research US, Inc. /ID# 210237, Greer, South Carolina
  - DeGarmo Institute of Medical Research /ID# 170528, Greer, South Carolina
  - Self Medical Group - Advanced /ID# 170336, Hodges, South Carolina
  - Main Street Physician's Care - Waterway /ID# 210441, Little River, South Carolina
  - PMG Research of Charleston /ID# 170572, Mt. Pleasant, South Carolina
  - Palmetto Institute of Clinical Research, Inc. /ID# 170395, Pelzer, South Carolina
  - Palmetto Clinical Research /ID# 170524, Summerville, South Carolina
  - Monument Health Clinical Research /ID# 170576, Rapid City, South Dakota
  - Holston Medical Group (Seasons of Bristol) /ID# 170565, Bristol, Tennessee
  - University Diabetes & Endocrine Consultants /ID# 170392, Chattanooga, Tennessee
  - Collierville Medical Specialists /ID# 170328, Collierville, Tennessee
  - PMG Research of Knoxville /ID# 170393, Jefferson City, Tennessee
  - Holston Medical Group Clinical /ID# 168165, Kingsport, Tennessee
  - New Phase Research & Development /ID# 170526, Knoxville, Tennessee
  - PMG Research of Knoxville /ID# 170451, Knoxville, Tennessee
  - PMG Research of Knoxville /ID# 170514, Knoxville, Tennessee
  - Baptist Memorial Medical Group Endocrine Clinic /ID# 168061, Memphis, Tennessee
  - Clinical Neuroscience Solutions - Memphis /ID# 170559, Memphis, Tennessee
  - Methodist Medical Group /ID# 168148, Memphis, Tennessee
  - University of Tennessee Health /ID# 170321, Memphis, Tennessee
  - Trinity Clinical Research, LLC /ID# 170369, Tullahoma, Tennessee
  - Arlington Family Research Center, Inc /ID# 170366, Arlington, Texas
  - Premier Family Physicians /ID# 167946, Austin, Texas
  - DiscoveResearch, Inc. /ID# 170320, Beaumont, Texas
  - Pioneer Research Solutions, Inc. /ID# 168062, Beaumont, Texas
  - Family Medicine Associates of Texas, PA /ID# 167849, Carrollton, Texas
  - 3rd Coast Research Associates /ID# 203091, Corpus Christi, Texas
  - Veterans Affairs North Texas Health Care System /ID# 170325, Dallas, Texas
  - Urology Clinics of North Texas /ID# 203033, Dallas, Texas
  - North TX Endocrine Center /ID# 170552, Dallas, Texas
  - Synexus Clinical Research US, INC /ID# 170319, Dallas, Texas
  - Village Health Partners - Legacy Medical Village /ID# 170659, Frisco, Texas
  - San Gabriel Clinical Research /ID# 167929, Georgetown, Texas
  - East Texas Cardiology /ID# 170638, Houston, Texas
  - PrimeCare Medical Group /ID# 168146, Houston, Texas
  - Associates in Medicine, P.A. /ID# 170439, Houston, Texas
  - Michael E. DeBakey VA Medical Center /ID# 167598, Houston, Texas
  - Discovery MM Services, Inc - Katy /ID# 202958, Houston, Texas
  - Centex Studies, Inc. - Houston /ID# 170537, Houston, Texas
  - Discovery MM Services, Inc - Houston - Broadway St /ID# 170558, Houston, Texas
  - The Endocrine Center /ID# 170653, Houston, Texas
  - Texas Center for Drug Development, Inc. /ID# 170404, Houston, Texas
  - Village Medical-MCA /ID# 170443, Houston, Texas
  - Methodist Urology Associates /ID# 170575, Houston, Texas
  - Endocrine and Psychiatry Cente /ID# 170520, Houston, Texas
  - Pioneer Research Solutions - Houston /ID# 170379, Houston, Texas
  - Research Trials Worldwide /ID# 210694, Humble, Texas
  - Protenium Clinical Research /ID# 170397, Hurst, Texas
  - Texas Cardio Association of Ho /ID# 170494, Kingwood, Texas
  - FMC Science /ID# 170407, Lampasas, Texas
  - Centex Studies, Inc /ID# 203019, McAllen, Texas
  - Discovery MM Services, Inc. /ID# 170562, Missouri City, Texas
  - Hill Country Medical Assoc /ID# 170444, New Braunfels, Texas
  - DCT-AACT, LLC dba Discovery Clinical Trials /ID# 170394, Pflugerville, Texas
  - ClinRx Research, LLC /ID# 203067, Plano, Texas
  - DeLeon Research /ID# 210861, Plano, Texas
  - Research Across America /ID# 168229, Plano, Texas
  - Texas Diabetes and Endocrinology - South Austin /ID# 170517, Round Rock, Texas
  - South Texas Cardiovascular Consultants /ID# 203088, San Antonio, Texas
  - Synexus Research - San Antonio /ID# 202947, San Antonio, Texas
  - Covenant Clinical Research, PA /ID# 170564, San Antonio, Texas
  - Victorium Clinical Research /ID# 168112, San Antonio, Texas
  - Northeast Clinical Research of San Antonio, LLC /ID# 202951, San Antonio, Texas
  - Discovery Clinical Trials-San Antonio /ID# 200845, San Antonio, Texas
  - ALM VA Hospital /ID# 167973, San Antonio, Texas
  - Consano Clinical Research, LLC /ID# 167848, Shavano Park, Texas
  - Spring Family Practice Associates, PA /ID# 203470, Spring, Texas
  - Hillcroft Medical Clinic /ID# 170500, Sugar Land, Texas
  - Northwest Houston Clinical Research PLLC /ID# 168223, Tomball, Texas
  - Crossroads Clinical Research, /ID# 170372, Victoria, Texas
  - Hillcrest Clinics /ID# 202961, Waco, Texas
  - Physicians Research Options, L /ID# 170441, Draper, Utah
  - Tanner Clinic /ID# 168145, Layton, Utah
  - Wasatch Peak Family Practice / Synexus Clinical Research US, Inc. /ID# 210175, Layton, Utah
  - Synexus Clinical Research US, Inc. /ID# 168248, Murray, Utah
  - Advanced Research Institute - Ridgeline /ID# 170445, Ogden, Utah
  - Optimum Clinical Research /ID# 170322, Salt Lake City, Utah
  - Velocity Clinical Research - Salt Lake City /ID# 167596, West Jordan, Utah
  - Connecticut Clinical Research Center /ID# 207771, Middlebury (village), Vermont
  - Burke Internal Medicine & Research /ID# 202981, Burke, Virginia
  - Seven Corners Medical Center /ID# 170577, Falls Church, Virginia
  - Manassas Clinical Research Center /ID# 201815, Manassas, Virginia
  - Virginia Research Center /ID# 170471, Midlothian, Virginia
  - Health Research of Hampton Roads, Inc. (HRHR) /ID# 204937, Newport News, Virginia
  - Clinical Research Associates of Tidewater /ID# 170609, Norfolk, Virginia
  - Clinical Research Partners LLC - Richmond Forest Ave /ID# 170490, Richmond, Virginia
  - Hunter Holmes McGuire VA Medical Center /ID# 170630, Richmond, Virginia
  - Salem VA Medical Center /ID# 167925, Salem, Virginia
  - Northwest Clinical Research Center /ID# 201588, Bellevue, Washington
  - Sound Medical Research /ID# 202938, Port Orchard, Washington
  - VA Puget Sound Health Care System /ID# 170555, Seattle, Washington
  - Universal Research Group, LLC /ID# 170442, Tacoma, Washington
  - American Health Network of Indiana, LLC /ID# 202987, Greenfield, Wisconsin
- Puerto Rico (5):
  - Emanuelli Research & Development Center LLC /ID# 206202, Arecibo
  - Research & Cardiovascular Corp /ID# 170353, Ponce
  - GCM Medical Group PSC /ID# 170466, San Juan
  - Centro de Endocrinologia Alcantara-Gonzalez /ID# 207260, San Juan
  - Advanced Clinical Research /ID# 170553, Toa Baja

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gagliano-Juca T, Pencina KM, Shang YV, Travison TG, Lincoff AM, Nissen SE, Artz AS, Li X, Chan A, Patel R, Miller MG, Bhasin S. Association of testosterone-induced increase in neutrophil and monocyte counts with thromboembolic events: The TRAVERSE trial. Am Heart J. 2025 Oct;288:77-88. doi: 10.1016/j.ahj.2025.04.004. Epub 2025 Apr 15. PMID 40246046
- [Derived] Bhasin S, Lincoff AM, Nissen SE, Wannemuehler K, McDonnell ME, Peters AL, Khan N, Snabes MC, Li X, Li G, Buhr K, Pencina KM, Travison TG. Effect of Testosterone on Progression From Prediabetes to Diabetes in Men With Hypogonadism: A Substudy of the TRAVERSE Randomized Clinical Trial. JAMA Intern Med. 2024 Apr 1;184(4):353-362. doi: 10.1001/jamainternmed.2023.7862. PMID 38315466
- [Derived] Snyder PJ, Bauer DC, Ellenberg SS, Cauley JA, Buhr KA, Bhasin S, Miller MG, Khan NS, Li X, Nissen SE. Testosterone Treatment and Fractures in Men with Hypogonadism. N Engl J Med. 2024 Jan 18;390(3):203-211. doi: 10.1056/NEJMoa2308836. PMID 38231621
- [Derived] Bhasin S, Travison TG, Pencina KM, O'Leary M, Cunningham GR, Lincoff AM, Nissen SE, Lucia MS, Preston MA, Khera M, Khan N, Snabes MC, Li X, Tangen CM, Buhr KA, Thompson IM Jr. Prostate Safety Events During Testosterone Replacement Therapy in Men With Hypogonadism: A Randomized Clinical Trial. JAMA Netw Open. 2023 Dec 1;6(12):e2348692. doi: 10.1001/jamanetworkopen.2023.48692. PMID 38150256
- [Derived] Pencina KM, Travison TG, Artz AS, Lincoff AM, Nissen SE, Flevaris P, Chan A, Li X, Diegel SA, Wannemuehler K, Bhasin S. Efficacy of Testosterone Replacement Therapy in Correcting Anemia in Men With Hypogonadism: A Randomized Clinical Trial. JAMA Netw Open. 2023 Oct 2;6(10):e2340030. doi: 10.1001/jamanetworkopen.2023.40030. PMID 37889486
- [Derived] Lincoff AM, Bhasin S, Flevaris P, Mitchell LM, Basaria S, Boden WE, Cunningham GR, Granger CB, Khera M, Thompson IM Jr, Wang Q, Wolski K, Davey D, Kalahasti V, Khan N, Miller MG, Snabes MC, Chan A, Dubcenco E, Li X, Yi T, Huang B, Pencina KM, Travison TG, Nissen SE; TRAVERSE Study Investigators. Cardiovascular Safety of Testosterone-Replacement Therapy. N Engl J Med. 2023 Jul 13;389(2):107-117. doi: 10.1056/NEJMoa2215025. Epub 2023 Jun 16. PMID 37326322
- See also: Related Info — http://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in the study across 316 sites in the US and Puerto Rico.
Pre-assignment Details: Of the 5246 participants randomized in the study, 42 participant identification numbers (IDs; AndroGel: 22 IDs; Placebo: 20 IDs) were randomized to 20 unique participants and these 42 duplicate/triplicate IDs were excluded from the Full Analysis Set. Additionally, a total of 6 randomized participants (AndroGel: 5 participants; Placebo: 1 participant) did not receive treatment and were excluded from the from the Safety Analysis Set, which resulted in 5198 participants in the Safety Analysis Set.
Groups:
- AndroGel 1.62%: Participants received topical testosterone starting with a 40.5 mg dose (2 pump actuations) of the study drug once daily (OD). Participants may have received a dose in the range of 20.25 mg (1 actuation) to 101.25 mg (5 actuations) in 20.25 mg increments during the course of the study if titrations were necessary.
- Placebo: Participants received matching placebo OD.
Period: Overall Study
Arm/Group | AndroGel 1.62% | Placebo
Started (Participants in Full Analysis Set (randomized, and no duplicate/triplicate participant IDs)) | 2601 | 2603
Participants in Safety Analysis Set (Randomized, Treated, no Duplicate/Triplicate Participant IDs) | 2596 | 2602
Completed | 1594 | 1581
Not Completed | 1007 | 1022
Not completed — Not Treated | 5 | 1
Not completed — Withdrawal by Subject | 309 | 351
Not completed — Lost to Follow-up | 446 | 458
Not completed — Adverse Event | 138 | 130
Not completed — Lack of Efficacy | 11 | 23
Not completed — COVID-19 Logistical Restriction | 7 | 3
Not completed — Serum Testosterone Level >750 ng/dL | 5 | 0
Not completed — Other, Not Specified | 84 | 53
Not completed — Reason Missing | 2 | 3

BASELINE CHARACTERISTICS:
Population: TRAVERSE Main Study Safety Set: All participants randomized with no duplicates who received at least one dose of study drug, grouped according to actual treatment received.
Groups:
- AndroGel 1.62%: Participants received topical testosterone starting with a 40.5 mg dose (2 pump actuations) of the study drug OD. Participants may have received a dose in the range of 20.25 mg (1 actuation) to 101.25 mg (5 actuations) in 20.25 mg increments during the course of the study if titrations were necessary.
- Total: Total of all reporting groups
Arm/Group | AndroGel 1.62% | Placebo | Total
Number analyzed (Participants) | 2596 | 2602 | 5198
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (7.93) | 63.3 (7.85) | 63.3 (7.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2596 | 2602 | 5198
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 409 | 439 | 848
  Not Hispanic or Latino | 2186 | 2161 | 4347
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 16 | 14 | 30
  Asian | 40 | 47 | 87
  Native Hawaiian or Other Pacific Islander | 14 | 7 | 21
  Black or African American | 445 | 432 | 877
  White | 2066 | 2083 | 4149
  More than one race | 15 | 18 | 33
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomization to the First Component Event of Major Adverse Cardiac Event (MACE): Number and Percentage of Participants With an Event
Description: MACE is a composite endpoint including non-fatal myocardial infraction (MI), non-fatal stroke and cardiovascular (CV) death as adjudicated by Clinical Events Committee (CEC).
Time Frame: Randomization to event or last known date if no event (up to approximately 52 months)
Population: TRAVERSE Main Study Safety Set: all randomized participants who received at least one dose of study drug and have no duplicate/triplicate participant IDs.
Measure: Count of Participants; unit: Participants
Arm/Group | AndroGel 1.62% | Placebo
Number analyzed (Participants) | 2596 | 2602
Participants | 182 | 190

2. Primary Outcome: Time From Randomization to the First Component Event of MACE
Description: MACE is a composite endpoint including non-fatal MI, non-fatal stroke and CV death as adjudicated by CEC.
Time Frame: Randomization to event or last known date if no event (up to approximately 52 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AndroGel 1.62% | Placebo
Number analyzed (Participants) | 2596 | 2602
months | NA [NA to NA] — Median and 95% confidence interval (CI) could not be calculated due to an insufficient number of events. | NA [NA to NA] — Median and 95% confidence interval (CI) could not be calculated due to an insufficient number of events.
Statistical Analysis 1: Comparison: AndroGel 1.62% vs Placebo; The hazard ratio (HR) and 2-sided 95% confidence interval (CI) were calculated using a Cox proportional-hazards regression model, with adjustment for pre-existing cardiovascular disease (CVD) status. In this analysis, the time to event for a participant is defined as the time from randomization to the first component event of MACE. If a subject does not experience a MACE during the study, the time is right-censored at the time of participant's last available follow-up observation; Test type: Non-Inferiority — Noninferiority margin in terms of HR is 1.5; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.78 to 1.17] — HR of AndroGel to placebo and 95% CI were estimated from Cox proportional-hazards regression model, with adjustment for pre-existing CVD

3. Secondary Outcome: Time From Randomization to the First Component Event of CV Safety Endpoint: Number and Percentage of Participants With an Event
Description: The CV safety endpoint is a composite endpoint including non-fatal MI, non-fatal stroke, CV death, and coronary revascularization procedures/cardiac percutaneous coronary intervention (PCI), or coronary artery bypass graft (CABG) as adjudicated by CEC.
Time Frame: Randomization to event or last known date if no event (up to approximately 52 months).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AndroGel 1.62% | Placebo
Number analyzed (Participants) | 2596 | 2602
Participants | 269 | 264

4. Secondary Outcome: Time From Randomization to the First Component Event of CV Safety Endpoint
Description: The CV safety endpoint is a composite endpoint including non-fatal MI, non-fatal stroke, CV death, and coronary revascularization procedures/cardiac PCI, or CABG as adjudicated by CEC.
Time Frame: Randomization to event or last known date if no event (up to approximately 52 months).
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AndroGel 1.62% | Placebo
Number analyzed (Participants) | 2596 | 2602
months | NA [NA to NA] — Median and 95% CI could not be calculated due to an insufficient number of events. | NA [NA to NA] — Median and 95% CI could not be calculated due to an insufficient number of events.
Statistical Analysis 1: Comparison: AndroGel 1.62% vs Placebo; The HR and 2-sided 95% CI were calculated using a Cox proportional-hazards regression model, with adjustment for pre-existing CVD status. In this analysis, the time to event for a participant is defined as the time from randomization to the first component event of CV safety endpoint. If a participant does not experience a CV safety endpoint during the study, the time is right-censored at the time of participant's last available follow-up observation; Test type: Superiority; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.86 to 1.21] — HR of AndroGel to placebo and 2-sided 95% CI were estimated from a Cox proportional-hazards regression model with adjustment of pre-existing CVD status

5. Secondary Outcome: Incidence of High-Grade Prostate Cancer
Description: Presented as the number and percentage of participants with any high grade prostate cancer, defined as Gleason grade of 4 + 3 or higher, as adjudicated by Prostate Safety Events Committee (PAC). This grade is based on how abnormal prostate cells appear. Grade 1: cells look almost like normal prostate cells; Grade 5; cells look very different from normal prostate cells. Since most prostate cancers contain cells of different grades, the 2 most common grades are used. Gleason score is determined by adding the 2 most common grades. Higher numbers indicate a faster growing cancer that is more likely to spread. Currently the lowest score assigned to a tumor is grade 3. Grades below 3 show normal to near normal cells. Most cancers have a Gleason score (the sum of the 2 most common grades) of 6 (Gleason scores of 3+3) or 7 (Gleason scores of 3+4 or 4+3).
Time Frame: Randomization to event or last known date if no event (up to approximately 52 months).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AndroGel 1.62% | Placebo
Number analyzed (Participants) | 2596 | 2602
Participants | 5 | 3
Statistical Analysis 1: Comparison: AndroGel 1.62% vs Placebo; The high grade prostate cancer endpoint was analyzed using a discrete time proportional hazard regression model with event time intervals based on scheduled visits, and adjusting for pre-existing CVD status. The HR of AndroGel to Placebo and its 2-sided 95% CI were provided; Test type: Superiority; Hazard Ratio (HR) = 1.62, 95% CI 2-sided [0.39 to 6.77] — Discrete-time proportional hazards model with event time intervals based on scheduled visits, and adjusting for prior cardiovascular disease (CVD)

6. Other Pre Specified Outcome: Change in Psychosexual Daily Questionnaire Question 4 (PDQ-Q4) From Baseline to Months 6, 12 and 24
Description: PDQ-Q4 asks 12 yes/no questions about sexual activity. Scores on the PDQ-Q4 range from 0 to 12, with higher scores indicating more activity.
Time Frame: From Baseline to Months 6, 12, and 24
Population: TRAVERSE Sexual Function Sub-Study: participants in the TRAVERSE main study full analysis set (i.e., randomized, no duplicate/triplicate participant IDs) who were eligible for the sexual function sub-study.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AndroGel 1.62% | Placebo
Number analyzed (Participants) | 260 | 259
score on a scale
  Change at Month 6 | 1.03 [0.82 to 1.24] | 0.54 [0.32 to 0.75]
  Change at Month 12: number analyzed (Participants) | 170 | 171
  Change at Month 12 | 0.97 [0.72 to 1.23] | 0.50 [0.25 to 0.76]
  Change at Month 24: number analyzed (Participants) | 106 | 95
  Change at Month 24 | 0.94 [0.60 to 1.28] | 0.46 [0.11 to 0.82]
Statistical Analysis 1: Comparison: AndroGel 1.62% vs Placebo; A linear mixed regression model was used to analyze the change in PDQ-Q4 from baseline to months 6, 12, and 24, with the dependent variable being the change in PDQ-Q4 score. The model included fixed effects for treatment, visit, and the interaction between treatment and visit, while adjusting for baseline PDQ-Q4 score and pre-existing CVD status. An unstructured covariance matrix was used to account for correlations among repeated measures within-subject; Test type: Superiority; p = 0.011, linear mixed regression model — P-value is derived from the omnibus likelihood-ratio chi-square test of the current model versus the null (intercept) model using linear mixed regression model; Omnibus likelihood-ratio chi-square test from linear mixed regression model
Statistical Analysis 2: Comparison: AndroGel 1.62% vs Placebo; Month 6 (results were derived from a linear mixed regression model that had a dependent variable of the change in PDQ-Q4 from baseline to months 6, 12, and 24. The model included fixed effects for treatment, visit, and the interaction between treatment and visit, while adjusting for baseline PDQ-Q4 score and pre-existing CV disease status. Additionally, an unstructured covariance matrix was used to account for correlations among repeated measures within participants); Test type: Superiority; LS Mean of Difference = 0.49, 95% CI 2-sided [0.19 to 0.79] — LS mean difference (AndroGel - Placebo) at month 6 was derived from linear mixed regression model
Statistical Analysis 3: Comparison: AndroGel 1.62% vs Placebo; Month 12 (results were derived from a linear mixed regression model that had a dependent variable of the change in PDQ-Q4 from baseline to months 6, 12, and 24. The model included fixed effects for treatment, visit, and the interaction between treatment and visit, while adjusting for baseline PDQ-Q4 score and pre-existing CV disease status. Additionally, an unstructured covariance matrix was used to account for correlations among repeated measures within participants); Test type: Superiority; LS Mean of Difference = 0.47, 95% CI 2-sided [0.11 to 0.83] — LS mean difference (AndroGel - Placebo) at month 12 was derived from linear mixed regression model
Statistical Analysis 4: Comparison: AndroGel 1.62% vs Placebo; Month 24 (results were derived from a linear mixed regression model that had a dependent variable of the change in PDQ-Q4 from baseline to months 6, 12, and 24. The model included fixed effects for treatment, visit, and the interaction between treatment and visit, while adjusting for baseline PDQ-Q4 score and pre-existing CV disease status. Additionally, an unstructured covariance matrix was used to account for correlations among repeated measures within participants); Test type: Superiority; LS Mean of Difference = 0.48, 95% CI 2-sided [-0.01 to 0.96] — LS mean difference (AndroGel - Placebo) at month 24 was derived from linear mixed regression model

7. Other Pre Specified Outcome: Number and Percentage of Participants Whose Persistent Depressive Disorder (PDD) Remits During Intervention Per Remission Definition
Description: The remission of low-grade, late-onset PDD was defined as: a) Patient Health Questionnaire (PHQ-9) score less than 4 and Geriatric Depression Scale-15 (GDS-15) score <5, and b) answer "no" to the question "Give your best guess: Over the past 6 months, have you been feeling sad or depressed more days than not, even if you felt okay sometimes?" The PHQ-9 is a 9-item depression scale. Total scores can range from 0 to 27, with higher scores indicating a worse outcome. A total score of 0-4 indicates minimal depression severity. The GDS-15 is a series of 15 yes/no questions asking how the participant felt in the past week. A score greater that 5 indicates depression; a higher score indicates a worse outcome.
Time Frame: Months 6, 12, 24
Population: PDD Sub-Study participants (those included TRAVERSE main study full analysis set participants [i.e., randomized, no duplicate/triplicate participant IDs] who met the criteria for low-grade PDD) with an assessment at given time point.
Measure: Count of Participants; unit: Participants
Arm/Group | AndroGel 1.62% | Placebo
Number analyzed (Participants) | 17 | 17
Participants
  Month 6 | 12 | 6
  Month 12: number analyzed (Participants) | 11 | 12
  Month 12 | 7 | 5
  Month 24: number analyzed (Participants) | 8 | 8
  Month 24 | 5 | 5
Statistical Analysis 1: Comparison: AndroGel 1.62% vs Placebo; Month 6 risk ratio of remission of LG-PDD in the AndroGel versus placebo group was estimated by a repeated measures generalized estimating equations (GEE) Poisson regression model with fixed effects for treatment, visit, treatment-visit interaction, pre- existing CVD, and an unstructured working correlation matrix to account for repeated measures at multiple visits; Test type: Superiority; Risk Ratio (RR) = 1.92, 95% CI 2-sided [0.96 to 3.86]
Statistical Analysis 2: Comparison: AndroGel 1.62% vs Placebo; Month 12 risk ratio of remission of LG-PDD in the AndroGel versus placebo group was estimated by a repeated measures generalized estimating equations (GEE) Poisson regression model with fixed effects for treatment, visit, treatment-visit interaction, pre- existing CVD, and an unstructured working correlation matrix to account for repeated measures at multiple visits; Test type: Superiority; Risk Ratio (RR) = 1.52, 95% CI 2-sided [0.64 to 3.63]
Statistical Analysis 3: Comparison: AndroGel 1.62% vs Placebo; Month 24 risk ratio of remission of LG-PDD in the AndroGel versus placebo group was estimated by a repeated measures generalized estimating equations (GEE) Poisson regression model with fixed effects for treatment, visit, treatment-visit interaction, pre- existing CVD, and an unstructured working correlation matrix to account for repeated measures at multiple visits; Test type: Superiority; Risk Ratio (RR) = 0.90, 95% CI 2-sided [0.42 to 1.94]
Statistical Analysis 4: Comparison: AndroGel 1.62% vs Placebo; Risk ratio of remission of LG-PDD in the TRT versus placebo group was estimated by a repeated measures generalized estimating equations (GEE) Poisson regression model with fixed effects for treatment, visit, treatment-visit interaction, pre- existing CVD, and an unstructured working correlation matrix to account for repeated measures at multiple visits; Test type: Superiority; p = 0.197, GEE Poisson regression model — The omnibus test p value is a test of the null hypothesis of no difference between AndroGel and placebo groups across all time points

8. Other Pre Specified Outcome: Time From Randomization to First Clinical Fracture: Number and Percentage of Participants With an Event
Description: Clinical fracture is defined as a clinical spine or non-spine fracture, documented by imaging or surgery, and confirmed by the Fracture Adjudication Committee (FAC). Fractures of the sternum, fingers, toes, facial bones and skull were excluded.
Time Frame: Randomization to event or last known date if no event (up to approximately 52 months).
Population: TRAVERSE Main Study Full Analysis Set: all randomized participants without duplicate/triplicate participant IDs.
Measure: Count of Participants; unit: Participants
Arm/Group | AndroGel 1.62% | Placebo
Number analyzed (Participants) | 2601 | 2603
Participants | 91 | 64

9. Other Pre Specified Outcome: Time From Randomization to First Clinical Fracture
Description: Clinical fracture is defined as a clinical spine or non-spine fracture, documented by imaging or surgery, and confirmed by the FAC. Fractures of the sternum, fingers, toes, facial bones and skull were excluded.
Time Frame: Randomization to event or maximum follow-up (up to approximately 52 months).
Population: TRAVERSE Main Study Full Analysis Set: all randomized participants without duplicate/triplicate participant IDs.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AndroGel 1.62% | Placebo
Number analyzed (Participants) | 2601 | 2603
months | NA [NA to NA] — Median and 95% CI could not be calculated due to an insufficient number of events. | NA [NA to NA] — Median and 95% CI could not be calculated due to an insufficient number of events.
Statistical Analysis 1: Comparison: AndroGel 1.62% vs Placebo; The HR and 2-sided 95% CI were calculated using a Cox proportional-hazards regression model, with adjustment for pre-existing CVD status. In this analysis, the time to event for a subject is defined as the time from randomization to the first occurrence of a clinical fracture. If a subject does not experience a clinic fracture during the study, the follow-up time is right-censored at the time of subject's last available follow-up observation; Test type: Superiority; Hazard Ratio (HR) = 1.43, 95% CI 2-sided [1.04 to 1.97] — Cox proportional-hazards model

10. Other Pre Specified Outcome: Number and Percentage of Anemic Participants Whose Baseline Anemia Was Corrected During the Intervention Period
Description: The correction of anemia was defined as an increase in hemoglobin level >12.7 g/dL during the intervention period (at Months 6, 12, 24, 36 and 48) for participants in TRAVERSE main study with anemia at baseline.
Time Frame: Baseline, Months 6, 12, 24, 36 and 48
Population: All randomized participants in TRAVERSE main study who had anemia at baseline; participants with an assessment at given time point.
Measure: Count of Participants; unit: Participants
Arm/Group | AndroGel 1.62% | Placebo
Number analyzed (Participants) | 349 | 375
Participants
  Month 6 | 143 | 103
  Month 12: number analyzed (Participants) | 338 | 360
  Month 12 | 152 | 122
  Month 24: number analyzed (Participants) | 290 | 307
  Month 24 | 124 | 95
  Month 36: number analyzed (Participants) | 216 | 229
  Month 36 | 94 | 76
  Month 48: number analyzed (Participants) | 92 | 97
  Month 48 | 41 | 38
Statistical Analysis 1: Comparison: AndroGel 1.62% vs Placebo; Repeated measures log-binomial regression with effects for treatment, visit, treatment-by-visit interaction, and adjusted for pre-existing CVD, and an unstructured covariance matrix to account for correlations among repeated measures within-subject; Test type: Other; p = 0.002, omnibus likelihood-ratio chi-square test — p-value is from an omnibus likelihood-ratio chi-square test of the current model versus the null (intercept) model using repeated measure log-binomial regression

11. Other Pre Specified Outcome: Number and Percentage of Participants With Pre-Diabetes at Baseline Who Progressed to Diabetes at Months 6, 12, 24, 36 and 48
Description: Number and percentage of participants in each arm who had prediabetes at baseline progressing to diabetes, defined as hemoglobin A1C (HbA1C) equal to or higher than 6.5%, initiation of diabetes medication, or two consecutive fasting glucose levels >125 mg/dL, assessed at all available time points after baseline.
Time Frame: Baseline, Months 6, 12, 24, 36 and 48
Population: All randomized participants in TRAVERSE main study who had prediabetes at baseline; participants with an assessment at given time point.
Measure: Count of Participants; unit: Participants
Arm/Group | AndroGel 1.62% | Placebo
Number analyzed (Participants) | 598 | 562
Participants
  Month 6 | 4 | 8
  Month 12: number analyzed (Participants) | 575 | 533
  Month 12 | 45 | 57
  Month 24: number analyzed (Participants) | 494 | 460
  Month 24 | 50 | 67
  Month 36: number analyzed (Participants) | 359 | 330
  Month 36 | 46 | 52
  Month 48: number analyzed (Participants) | 164 | 121
  Month 48 | 22 | 19
Statistical Analysis 1: Comparison: AndroGel 1.62% vs Placebo; The risk ratio of progression to diabetes in the AndroGel versus placebo group was estimated by a repeated measures log-binomial regression with fixed effects for treatment, visit, treatment-visit interaction, and pre-existing CVD, and an unstructured covariance matrix to account for correlations among repeated measures within-subject; Test type: Superiority; p = 0.494, Repeated measures log-binomial regr. — [p-value comment as in outcome 10, analysis 1]

12. Other Pre Specified Outcome: Tertiary Endpoint: Incidence Rate of All Cause Mortality
Description: Presented as the number and percentage of participants who died, regardless of cause.
Time Frame: Randomization to event or last known date if no date (up to approximately 52 months).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AndroGel 1.62% | Placebo
Number analyzed (Participants) | 2596 | 2602
Participants | 144 | 148
Statistical Analysis 1: Comparison: AndroGel 1.62% vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.78 to 1.23] — Cox proportional-hazards model adjusting for prior CVD

13. Other Pre Specified Outcome: Tertiary Endpoint: Incidence Rate of Heart Failure
Description: Presented as the number and percentage of participants with heart failure events (requiring hospitalization and/or urgent visit), as adjudicated by CEC.
Time Frame: Randomization to event or last known date if no date (up to approximately 52 months).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AndroGel 1.62% | Placebo
Number analyzed (Participants) | 2596 | 2602
Participants | 55 | 50
Statistical Analysis 1: Comparison: AndroGel 1.62% vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.76 to 1.62] — Cox proportional-hazards model adjusting for prior CVD

14. Other Pre Specified Outcome: Tertiary Endpoint: Incidence Rate of Venous Thromboembolic Events
Description: Presented as the number and percentage of participants with venous thromboembolic events, as adjudicated by CEC. Events include deep vein thrombosis, pulmonary embolism, venous thromboembolism (excluding superficial thrombophlebitis).
Time Frame: Randomization to event or last known date if no date (up to approximately 52 months).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AndroGel 1.62% | Placebo
Number analyzed (Participants) | 2596 | 2602
Participants | 44 | 30
Statistical Analysis 1: Comparison: AndroGel 1.62% vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.46, 95% CI 2-sided [0.92 to 2.32] — Cox proportional-hazards model adjusting for prior CVD

15. Other Pre Specified Outcome: Tertiary Endpoint: Incidence Rate of Peripheral Arterial Revascularization
Description: Presented as the number and percentage of participants with peripheral arterial revascularization, as adjudicated by CEC.
Time Frame: Randomization to event or last known date if no event (up to approximately 52 months).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AndroGel 1.62% | Placebo
Number analyzed (Participants) | 2596 | 2602
Participants | 30 | 33
Statistical Analysis 1: Comparison: AndroGel 1.62% vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.56 to 1.51] — Cox proportional-hazards model adjusting for prior CVD

16. Other Pre Specified Outcome: Tertiary Endpoint: Incidence Rate of Prostate Biopsy
Description: Presented as the number and percentage of participants who underwent prostate biopsy.
Time Frame: Randomization to event or last known date if no event (up to approximately 52 months).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AndroGel 1.62% | Placebo
Number analyzed (Participants) | 2596 | 2602
Participants | 16 | 14
Statistical Analysis 1: Comparison: AndroGel 1.62% vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.55 to 2.31] — Discrete-time proportional hazards model with event time intervals based on scheduled visits, and adjusting for prior CVD

17. Other Pre Specified Outcome: Tertiary Endpoint: Incidence Rate of Prostate Cancer
Description: Presented as the number and percentage of participants who with prostate cancer, as adjudicated by Prostate Safety Events Committee (PAC).
Time Frame: Randomization to event or last known date if no event (up to approximately 52 months).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AndroGel 1.62% | Placebo
Number analyzed (Participants) | 2596 | 2602
Participants | 12 | 11
Statistical Analysis 1: Comparison: AndroGel 1.62% vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.47 to 2.42] — [estimate comment as in outcome 16, analysis 1]

18. Other Pre Specified Outcome: Tertiary Endpoint: Incidence Rate of Acute Urinary Retention
Description: Presented as the number and percentage of participants with acute urinary retention, as adjudicated by PAC.
Time Frame: Randomization to event or last known date if no event (up to approximately 52 months).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AndroGel 1.62% | Placebo
Number analyzed (Participants) | 2596 | 2602
Participants | 20 | 16
Statistical Analysis 1: Comparison: AndroGel 1.62% vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [0.65 to 2.41] — [estimate comment as in outcome 16, analysis 1]

19. Other Pre Specified Outcome: Tertiary Endpoint: Incidence Rate of Pharmacologic Treatment for Lower Urinary Tract Symptoms
Description: Presented as the number and percentage of participants who started pharmacologic treatment for lower urinary tract symptoms.
Time Frame: Randomization to event or last known date if no event (up to approximately 52 months).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AndroGel 1.62% | Placebo
Number analyzed (Participants) | 2596 | 2602
Participants | 101 | 87
Statistical Analysis 1: Comparison: AndroGel 1.62% vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.87 to 1.54] — [estimate comment as in outcome 16, analysis 1]

20. Other Pre Specified Outcome: Tertiary Endpoint: Incidence Rate of Invasive Prostate Surgical Procedures for Benign Prostatic Hyperplasia
Description: Presented as the number and percentage of participants who underwent invasive prostate surgical procedures for benign prostate hyperplasia, as adjudicated by Prostate Safety Events Committee (PAC). Invasive prostate surgical procedures include prostatectomy, transurethral prostate resection, brachytherapy or other prostate surgical procedure.
Time Frame: Randomization to event or last known date if no event (up to approximately 52 months).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AndroGel 1.62% | Placebo
Number analyzed (Participants) | 2596 | 2602
Participants | 23 | 12
Statistical Analysis 1: Comparison: AndroGel 1.62% vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.91, 95% CI 2-sided [0.95 to 3.84] — [estimate comment as in outcome 16, analysis 1]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs): from enrollment to 30 days post last dose (up to Month 48). Non-serious adverse events (AEs): from first dose of study drug to 30 days post last dose (up to Month 48). All-cause mortality (ACM): entire study duration (up to approximately 52 months).
Description: Other AEs were not collected prior to first dose, per protocol.
Groups:
- AndroGel 1.62% Predose: Participants randomized to the AndroGel 1.62% arm, prior to first dose.
- Placebo Predose: Participants randomized to the Placebo arm, prior to first dose.
Arm/Group | AndroGel 1.62% Predose | Placebo Predose | AndroGel 1.62% | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2601 | 0/2603 | 144/2601 | 148/2603
Serious Adverse Events (participants affected / at risk) | 19/2601 | 10/2603 | 585/2601 | 562/2603
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 160/2601 | 170/2603
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AndroGel 1.62% Predose (N=2601) | Placebo Predose (N=2603) | AndroGel 1.62% (N=2601) | Placebo (N=2603)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 7 (7) | 6 (7)
BLOOD LOSS ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
POLYCYTHAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
ACUTE LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 30 (31) | 30 (31)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0) | 10 (10) | 22 (23)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1) | 0 (0) | 19 (20) | 32 (35)
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
AORTIC VALVE STENOSIS (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 37 (40) | 30 (35)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 1 (1) | 9 (9) | 5 (5)
ATRIAL TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 1 (1) | 0 (0) | 8 (8) | 13 (14)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 5 (5) | 3 (5)
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 0 (0) | 0 (0) | 8 (8) | 6 (6)
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 0 (0) | 0 (0) | 10 (11) | 7 (7)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 13 (13) | 9 (9)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 6 (7) | 7 (8)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 (0) | 0 (0) | 14 (14) | 13 (13)
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 23 (29) | 25 (32)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
CARDIOGENIC SHOCK (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 6 (6)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIOVASCULAR DISORDER (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
CHRONIC LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1) | 32 (33) | 35 (40)
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 0 (0) | 0 (0) | 7 (7) | 4 (4)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 (0) | 0 (0) | 8 (8) | 0 (0)
DEFECT CONDUCTION INTRAVENTRICULAR (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENDOCARDITIS NONINFECTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSIVE HEART DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INTRACARDIAC THROMBUS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 24 (25) | 21 (21)
MYOCARDIAL INJURY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
PALPITATIONS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PERICARDITIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULSELESS ELECTRICAL ACTIVITY (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
SINUS ARRHYTHMIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 6 (6) | 11 (12)
SINUS NODE DYSFUNCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 7 (7) | 11 (11)
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 9 (9) | 4 (4)
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 9 (9) | 7 (8)
CEREBRAL CAVERNOUS MALFORMATION (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PHIMOSIS (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HYPERPARATHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
THYROID CYST (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLINDNESS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLINDNESS UNILATERAL (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIPLOPIA (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RETINAL ARTERY OCCLUSION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
VISION BLURRED (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VISUAL IMPAIRMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
ABDOMINAL WALL HAEMATOMA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASCITES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BARRETT'S OESOPHAGUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COLON DYSPLASIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
CROHN'S DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIVERTICULUM (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DUODENAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DUODENAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6) | 7 (8)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 3 (3)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOAESTHESIA ORAL (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OBSTRUCTIVE PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PANCREATIC MASS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 3 (3)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
PNEUMOPERITONEUM (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RECTAL FISSURE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
CARDIAC DEATH (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHEST DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
DEATH (General disorders) | 0 (0) | 0 (0) | 5 (5) | 8 (8)
DROWNING (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ELECTROCUTION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
HERNIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOTHERMIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
IMPAIRED HEALING (General disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
INFLAMMATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MEDICAL DEVICE PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 20 (21) | 16 (16)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ORGAN FAILURE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PAIN (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
PELVIC MASS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERIPHERAL SWELLING (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
SOFT TISSUE INFLAMMATION (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STENT-GRAFT ENDOLEAK (General disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
SUDDEN CARDIAC DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
TREATMENT NONCOMPLIANCE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UNEVALUABLE EVENT (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VASCULAR STENT OCCLUSION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VASCULAR STENT STENOSIS (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BILE DUCT STONE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BILIARY DYSKINESIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 5 (5) | 3 (4)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEPATIC MASS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONTRAST MEDIA ALLERGY (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
IMMUNISATION REACTION (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACINETOBACTER INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
APPENDICITIS PERFORATED (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ARTHRITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
ARTHRITIS INFECTIVE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ATYPICAL PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
CANDIDA SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 22 (24) | 35 (35)
CELLULITIS GANGRENOUS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CELLULITIS OF MALE EXTERNAL GENITAL ORGAN (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CELLULITIS STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CITROBACTER INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
CORONAVIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 38 (38) | 19 (19)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 27 (27) | 22 (22)
DEVICE RELATED BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
DIABETIC FOOT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 6 (6) | 4 (4)
EMPYEMA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
ENDOCARDITIS (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
ENDOCARDITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ENDOPHTHALMITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENTEROBACTER INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENTEROCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EPIDIDYMITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ERYSIPELAS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ESCHERICHIA SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
EXTRADURAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GANGRENE (Infections and infestations) | 0 (0) | 0 (0) | 6 (7) | 4 (4)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
HAEMATOMA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEPATITIS A (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 6 (6) | 3 (3)
INTERVERTEBRAL DISCITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
KLEBSIELLA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
KLEBSIELLA SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 9 (9)
MASTOIDITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MEDICAL DEVICE SITE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MENINGITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NECROTISING SOFT TISSUE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ORCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 0 (0) | 14 (18) | 15 (17)
OSTEOMYELITIS ACUTE (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PNEUMOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 37 (42) | 35 (37)
PNEUMONIA ASPIRATION (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA KLEBSIELLA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA LEGIONELLA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA PSEUDOMONAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
POST PROCEDURAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POST-ACUTE COVID-19 SYNDROME (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PROSTATIC ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PROTEUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PSEUDOMONAS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
RHINOVIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SCROTAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SCROTAL CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SCROTAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 2 (2) | 0 (0) | 20 (20) | 21 (21)
SEPSIS SYNDROME (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
SEPTIC CEREBRAL EMBOLISM (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SEPTIC ENCEPHALOPATHY (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 8 (8) | 4 (4)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
STAPHYLOCOCCAL OSTEOMYELITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
STREPTOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
SUBACUTE ENDOCARDITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
URETHRAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 8 (8)
UROSEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
ARTERIAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AVULSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COMMINUTED FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CRUSH INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
DEEP VEIN THROMBOSIS POSTOPERATIVE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIFFUSE AXONAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 5 (5) | 12 (12)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
FOREIGN BODY IN THROAT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FRACTURE DISPLACEMENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
HEAT STROKE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
IATROGENIC INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LIMB TRAUMATIC AMPUTATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OPEN FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
PERIPROSTHETIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
POSTOPERATIVE RESPIRATORY FAILURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POSTOPERATIVE THORACIC PROCEDURE COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
PULMONARY CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 4 (4) | 5 (5)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 8 (8) | 3 (3)
SCAPULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKIN ABRASION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKULL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
THIRD DEGREE CHEMICAL BURN OF SKIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
TRAUMATIC LIVER INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ULNA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VASCULAR GRAFT OCCLUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
WOUND (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
BLOOD PRESSURE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
BRAIN NATRIURETIC PEPTIDE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EJECTION FRACTION DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LIVER FUNCTION TEST INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PROCALCITONIN INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PROSTATIC SPECIFIC ANTIGEN INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SARS-COV-2 TEST NEGATIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TROPONIN INCREASED (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
JAW FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
STRESS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TRAUMATIC RENAL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SINUS RHYTHM (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 6 (6) | 3 (3)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (5) | 8 (8)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 6 (6)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
HYPERGLYCAEMIC HYPEROSMOLAR NONKETOTIC SYNDROME (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERVOLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 5 (6)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
KETOACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
OBESITY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
POLYDIPSIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (6) | 5 (5)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (6) | 4 (4)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NECK DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 14 (16) | 18 (18)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
POLYMYALGIA RHEUMATICA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
TEMPOROMANDIBULAR JOINT SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VERTEBRAL FORAMINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
CHEST WALL HAEMATOMA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ADENOCARCINOMA GASTRIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
ADENOCARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
BONE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARCINOID TUMOUR OF THE SMALL BOWEL (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHOLANGIOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CLEAR CELL RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COLORECTAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FOLLICULAR THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL STROMAL TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEPATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEPATIC CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HODGKIN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LARYNGEAL SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LIPOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
LUNG SQUAMOUS CELL CARCINOMA STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MALIGNANT ASCITES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MALIGNANT MELANOMA STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MANTLE CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MENINGIOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
METASTASES TO LYMPH NODES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MONOCLONAL GAMMOPATHY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEUROENDOCRINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
NON-SMALL CELL LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NON-SMALL CELL LUNG CANCER STAGE IIIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NON-SMALL CELL LUNG CANCER STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OROPHARYNGEAL SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PITUITARY TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PITUITARY TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PLASMA CELL MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
PLASMA CELL MYELOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 6 (6) | 7 (7)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RECTAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RECTAL CANCER STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
SALIVARY GLAND CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
THROAT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AMNESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
APHASIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
ATAXIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AUTONOMIC NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BELL'S PALSY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
BRAIN STEM HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (4)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CAUDA EQUINA SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CEREBELLAR INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CEREBELLAR STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CEREBRAL HAEMATOMA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CEREBRAL VENTRICLE DILATATION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 9 (9) | 13 (13)
CERVICAL CORD COMPRESSION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CERVICAL RADICULOPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
CLONIC CONVULSION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CRANIAL NERVE PARALYSIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIABETIC NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 6 (6) | 5 (5)
DYSARTHRIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
ESSENTIAL TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GUILLAIN-BARRE SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMORRHAGIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
HAEMORRHAGIC TRANSFORMATION STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HEMIPARESIS (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
HYPOXIC-ISCHAEMIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INTRACRANIAL HAEMATOMA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 12 (12) | 6 (6)
LACUNAR INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LACUNAR STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
LUMBAR RADICULOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
MENINGEAL THICKENING (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MYASTHENIA GRAVIS (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (4)
MYELOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NORMAL PRESSURE HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PARALYSIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 5 (5) | 5 (5)
QUADRIPARESIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RADIAL NERVE PALSY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
RADICULOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
SPEECH DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPINAL CLAUDICATION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 22 (27) | 22 (23)
THROMBOTIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TOXIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
TRANSIENT GLOBAL AMNESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 0 (0) | 6 (6) | 13 (13)
TRIGEMINAL NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SQUAMOUS CELL CARCINOMA OF HEAD AND NECK (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SPINAL EPIDURAL HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEVICE DISLOCATION (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEVICE FAILURE (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEVICE OCCLUSION (Product Issues) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
ADJUSTMENT DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AGGRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALCOHOL ABUSE (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
BIPOLAR II DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COMPLETED SUICIDE (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DELIRIUM (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
MAJOR DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
MANIA (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PANIC ATTACK (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERSONALITY DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POST-TRAUMATIC STRESS DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 0 (0) | 31 (31) | 25 (25)
CALCULUS BLADDER (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
CALCULUS URINARY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
END STAGE RENAL DISEASE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 5 (6) | 5 (5)
OBSTRUCTIVE NEPHROPATHY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
POLYURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RENAL COLIC (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
RENAL HAEMATOMA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RENAL HAEMORRHAGE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URETERIC OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
URETEROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
URETHRAL OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINARY BLADDER HERNIATION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 9 (9) | 9 (9)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PRIAPISM (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PROSTATOMEGALY (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 36 (39) | 24 (26)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRONCHIAL HYPERREACTIVITY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 13 (16) | 13 (14)
CHRONIC RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 8 (8) | 8 (8)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERCAPNIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 12 (13) | 2 (2)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OBSTRUCTIVE SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PHARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PNEUMOMEDIASTINUM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 17 (17) | 8 (8)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
PULMONARY FISTULA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 8 (8) | 6 (6)
TRACHEAL CALCIFICATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIABETIC FOOT (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
DIABETIC ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIABETIC WOUND (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 3 (3)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
IMMOBILE (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AMPUTATION (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANGIOPLASTY (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIAC PACEMAKER REPLACEMENT (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HIP ARTHROPLASTY (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
KNEE ARTHROPLASTY (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
LEG AMPUTATION (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPINAL FUSION SURGERY (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STENT PLACEMENT (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TOE AMPUTATION (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AORTIC ANEURYSM (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
AORTIC STENOSIS (Vascular disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
ARTERIAL HAEMORRHAGE (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ARTERIAL THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTERIOSCLEROSIS (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 8 (9) | 10 (10)
HAEMATOMA (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
HYPERTENSIVE CRISIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HYPERTENSIVE EMERGENCY (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
HYPERTENSIVE URGENCY (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 5 (5) | 8 (8)
ILIAC ARTERY STENOSIS (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
INTERMITTENT CLAUDICATION (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
MALIGNANT HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 (0) | 0 (0) | 5 (8) | 6 (8)
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERIPHERAL ARTERY OCCLUSION (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 0 (0) | 0 (0) | 5 (5) | 3 (3)
PERIPHERAL VENOUS DISEASE (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SHOCK HAEMORRHAGIC (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SUBCLAVIAN VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
VASCULAR COMPRESSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VASCULAR STENOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VENOUS THROMBOSIS LIMB (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | AndroGel 1.62% Predose (N=0) | Placebo Predose (N=0) | AndroGel 1.62% (N=2601) | Placebo (N=2603)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 160/2596 (169) | 170/2602 (183)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT03518034/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT03518034/SAP_001.pdf